CLINICAL TRIAL: NCT06682416
Title: The Impact of Local Anesthetic Solution Temperature on Epidural-related Maternal Fever
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Fuhai Ji, Director, department of anesthesiology, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023367
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Epidural Related Maternal Fever; Analgesia, Epidural; Fever; Intrapartum Fever
MeSH Terms: conditions — Agnosia; Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation group (Experimental): Participants will be assigned to receive 37°C local anesthetic solutions.
  Interventions: Procedure: In the context of epidural analgesia, the temperature of the local anesthetic solution is elevated to 37°C utilizing a blood transfusion and infusion warmer.
- Control group (No Intervention): Participants will be assigned to receive 23°C local anesthetic solutions.

INTERVENTIONS:
Procedure: In the context of epidural analgesia, the temperature of the local anesthetic solution is elevated to 37°C utilizing a blood transfusion and infusion warmer. — For the observation group, after reactivating the analgesic pump's exhaust procedure to clear the air from the tubing, the output tubing of the analgesic pump is first connected to the epidural catheter. Following this, a blood transfusion and infusion warmer (manufactured by Barkey GmbH & Co. KG., Germany, model S-line, with the national medical device registration number 20182450063) is used to preheat the output tubing of the analgesic pump until it reaches the predetermined temperature of 37°C.
  For the control group, after reactivating the analgesic pump's exhaust procedure to remove air from the tubing, the output tubing of the analgesic pump is connected to the epidural catheter without preheating the output tubing using a blood transfusion and infusion warmer, maintaining room temperature (23°C).
  Arms: Observation group

SUMMARY:
This study investigates how the temperature of local anesthetics affects maternal fever related to epidural analgesia during childbirth. The research is a prospective, randomized controlled trial involving 424 participants from two hospitals. The primary objective is to investigate the impact of local anesthetic solution temperature on intrapartum fever in parturients. Secondary goals include assessing the impact on the efficacy of epidural analgesia and various maternal and neonatal outcomes. Participants will receive either 37°C or 23°C anesthetic solutions, and data will be collected on fever rates, pain scores, and other health indicators. The study runs from January 2024 to December 2026.

DETAILED DESCRIPTION:
Background:

Maternal fever during labor is common, with an incidence of about 33%, often due to infection, epidural analgesia, or environmental factors. Multiple studies have indicated that the rate of intrapartum fever in women who receive epidural analgesia is approximately between 15% and 25%. After epidural analgesia, the risk of maternal fever significantly increases, a condition known as Epidural-Related Maternal Fever (ERMF). ERMF not only increases unnecessary antibiotic use but may also lead to unplanned cesarean sections, increased perinatal bleeding, and other complications. Moreover, any cause of intrapartum fever, including ERMF, can increase the incidence of neonatal brain injury by approximately 2.79 times. With the popularization of the concept of painless childbirth, ERMF has increasingly attracted people's attention. Despite being identified in 1989, the pathogenesis of ERMF remains unclear, with several mechanisms proposed, including infection, sympathetic blockade, and non-infectious inflammation induced by local anesthetics.

Methods:

This is a prospective randomized controlled study with 424 participants receiving epidural analgesia at two hospitals from October 2024 to October 2027. Participants will be randomly assigned to receive either 37°C or 23°C local anesthetic solutions. The study will measure maternal fever rates, the time for pain scores to decrease, and peripheral perfusion index at various intervals. Maternal and neonatal outcomes, including antibiotic usage, sepsis incidence, and Apgar scores, will be recorded.

Possible Conclusions:

The study aims to determine if the temperature of local anesthetics influences the incidence of ERMF. It also seeks to assess the impact of anesthetic temperature on the onset and duration of epidural analgesia and various maternal and neonatal health outcomes. The findings may provide evidence on whether warming local anesthetics can reduce the risk of ERMF and improve maternal and neonatal health during labor.

ELIGIBILITY:
Inclusion Criteria:

1. Requesting epidural analgesia;
2. Aged 18 or older;
3. At least 37 weeks of gestation;
4. Those delivering vaginally.

Exclusion Criteria:

1. Contraindications to epidural analgesia;
2. Pre-existing fever (≥38°C) before labor;
3. Use of NSAIDs or other types of antipyretics before labor;
4. Multiple pregnancy (carrying more than one fetus);
5. Fetal demise (stillbirth);
6. Severe preeclampsia;
7. Women who refuse to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Maternal fever incidence | Before epidural catheterization, and at 2, 4, and 6 hours after epidural catheterization, and at the end of the second and third stages of labor, and 1 hour postpartum.
  The primary outcome measure for this trial is the incidence of maternal fever, as determined by oral temperature readings, throughout the entire labor process. Maternal fever is defined as maternal intrapartum fever with a temperature of 38°C or higher.

SECONDARY OUTCOMES:
VAS ≤ 3 | From date of receiving epidural anesthesia until the date of VAS ≤ 3, an average of 30 minutes
  The Visual Analogue Scale (VAS) is a simple tool for assessing pain intensity. It features a 100mm line with "0" at one end indicating no pain and "10" at the other end representing the worst possible pain. Patients mark their pain level anywhere along the line, providing a continuous measure of their discomfort.
Pulse Perfusion Index | Before epidural anesthesia, and at 10 minutes, 20 minutes, and 30 minutes after epidural catheterization.
Maternal and Neonatal Antibiotic Use Rate | From the date of randomization until the date of first documented maternal or neonatal antibiotic use, assessed up to 1 month postoperatively.
  Querying the electronic medical record system for antibiotic usage
Incidence of bacteremia | From the date of randomization until the date of first documented bacteremia, assessed up to 1 month postoperatively.
  The proportion of positive bacterial culture test results in each group.
Intrapartum hypothermia | Before epidural catheterization, and at 2, 4, and 6 hours after epidural catheterization, and at the end of the second and third stages of labor, and 1 hour postpartum.
Duration of labor | From the onset of labor until the delivery of the placenta, assessed up to 48 hours.
Unplanned cesarean section rate | From date of randomization until the delivery of the placenta, assessed up to 48 hours.
Umbilical Artery pH | up to 48 hours
  After the delivery of the fetus, umbilical arterial blood is drawn to check the pH of the umbilical artery.
Apgar score at 1st and 5th minute for newborns | From the minute of fetal delivery until 5th minute post-delivery, assessed up to 5 minutes post-delivery.
  After the delivery of the fetus, the Apgar score is assessed at the 1st and 5th minute post-delivery. The Apgar score is a quick test used to assess the physical condition of a newborn baby immediately after birth. It is performed at one and five minutes after birth, and sometimes at 10 and 20 minutes as well. The score is based on five criteria: Appearance (skin color), Pulse (heart rate), Grimace (reflex irritability), Activity (muscle tone), and Respiration (breathing). Each category is scored on a scale from 0 to 2, with 0 indicating the worst condition and 2 the best. The total score ranges from 0 to 10, with a score of 7 to 10 generally considered normal, 4 to 6 indicating the need for some medical assistance, and below 4 requiring immediate medical attention.

CONTACTS AND LOCATIONS:
Overall Officials: Fuhai Ji, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (2):
- China (2):
  - Ethical Committee of the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
We will share the raw data on ResMan (www.medresman.org.cn). Additionally, the research data will be published in the form of a paper within 2 years after the completion of the clinical trial.

REFERENCES:
- [Derived] Chen D, Wang Q, Wu Q, Shen M, Zhang J, Shan X, Feng CD, Tang H, Wei L, Ji F. Body-temperature versus room-temperature local anaesthetic solutions for epidural-related maternal fever prevention in labour: protocol for a two-centre randomised controlled trial. BMJ Open. 2025 Nov 4;15(11):e101760. doi: 10.1136/bmjopen-2025-101760. PMID 41193197